CLINICAL TRIAL: NCT00996177
Title: Comparison of Transdermal Fentanyl PCA and IV Morphine PCA in the Management of Postoperative Pain Control
Brief Title: A Study to Compare Patient-controlled Pain Medications Delivered Either Through the Skin or Intravenously
Acronym: EuroTrans
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen-Cilag International NV (Industry)
Collaborators: Alza Corporation, DE, USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR003943; FEN-PPA-401 (Other: Janssen-Cilag International); 2004-001201-10 (EudraCT Number)
Record Dates: First submitted 2009-09-28; First posted 2009-10-16 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2014-01

CONDITIONS: Pain; Analgesia, Patient-Controlled; Pain, Postoperative
Keywords: Pain; Patient-controlled analgesia; Postoperative pain; Transdermal fentanyl; Surgical pain; Opioid analgesics
MeSH Terms: conditions — Pain; Agnosia; Pain, Postoperative | interventions — Fentanyl; Analgesia, Patient-Controlled

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IONSYS (Experimental): IONSYS (fentanyl HCl) Iontophoretic TransdermalSystem
  Interventions: Drug: IONSYS (fentanyl HCl) Iontophoretic TransdermalSystem
- Patient-Controlled Analgesia (Active Comparator): IV Morphine Patient-Controlled Analgesia (IV PCA)
  Interventions: Drug: IV Morphine Patient-Controlled Analgesia (IV PCA)

INTERVENTIONS:
Drug: IONSYS (fentanyl HCl) Iontophoretic TransdermalSystem — 40 µg fentanyl on-demand (240µg/hr) or a maximum of 80 doses (3.2 mg) per day
  Arms: IONSYS
Drug: IV Morphine Patient-Controlled Analgesia (IV PCA) — 20mg/2hr (240 mg during 24 hours)
  Arms: Patient-Controlled Analgesia

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of a patient-controlled system to deliver fentanyl compared with a patient-controlled intravenous system to deliver morphine in the management of postoperative pain.

DETAILED DESCRIPTION:
This is a randomized (study drug assigned by chance), open-label (all people involved know the identity of the intervention) study to evaluate the clinical use, safety and ease of care of two patient-controlled analgesia (PCA) systems to deliver pain medication either through the skin or intravenously. The fentanyl hydrochloride PCA system, which delivers the medication through the skin, and morphine intravenous (IV)- PCA, which requires injection into a vein, are used for management of moderate to severe acute pain in postoperative patients who have undergone elective major abdominal or orthopedic surgery. These patients, who are expected to require postoperative pain relief with strong opioids for at least 24 hours, will control the delivery of medication for up to 3 days. Assessment of effectiveness include: patient's global assessment of pain control (poor, fair, good, excellent); Pain Intensity, measured on a visual numerical rating scale from 0 to 10, where 0 means no pain and 10 means the worst possible pain; Ease-of-Care questionnaires including Patient Ease-of-Care questionnaire, Nurse Ease-of-Care questionnaire, and Physical Therapist Ease-of-Care questionnaire; and, total number of doses delivered by patients in the fentanyl transdermal PCA or morphine IV PCA treatment groups. Safety evaluations include vital signs (pulse, blood pressure) and oxygen saturation, respiratory function, and the incidence of adverse events. The study hypothesis is that fentanyl transdermal PCA is not inferior to morphine IV PCA treatment in patient's global assessment of method of pain control during the first 24 hours after surgery. Transdermal PCA: 40 micrograms fentanyl per on-demand dose, each delivered over 10 minutes for a maximum of 6 doses/hr for 24 hours (maximum of 80 doses, 3.2milligrams). Morphine IV PCA: morphine doses with a maximum of 20 milligrams per 2 hours for 24 hours (maximum 12 doses, 240 milligrams).

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet the criteria of American Society of Anesthesiology (ASA) pre-operative physical status I, II, or III
* Patients expected to have moderate or severe pain after a major abdominal or orthopedic procedure
* Patients expected to remain hospitalized for at least 24 hours postoperatively

Exclusion Criteria:

* Known allergy or hypersensitivity to fentanyl, morphine, or to skin adhesives
* Known or suspected to be dependent on strong opioids or to have abused any drug substance or alcohol
* Severe respiratory symptoms
* Chronic pain disorder
* Pregnant or nursing women, or those lacking adequate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 657 (Actual)
Dates: Start 2004-06; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Patient's global assessment of pain control (poor, fair, good, excellent) 24 hours after start of study treatment | 24 hours after randomization (24 hours after either the first transdermal iontorphoretic system was applied or 24 hours after the intravenous access for the morphine solution was applied).

SECONDARY OUTCOMES:
Assessment of pain control by patient and doctor | At 24, 48, and 72 hours after randomization
Pain Intensity, vital signs, and oxygen level in the blood | Hourly through 8 hours and then every 4 hours after randomization
Incidence of adverse events | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (44):
- Vienna, Austria
- Belgium (3):
  - Brussels
  - Ghent
  - Leuven
- Denmark (5):
  - Aalborg
  - Kÿbenhavn Nv N/A
  - Kÿbenhavn Ÿ
  - Odense C
  - Ÿrhus C
- France (8):
  - Boulogne-Billancourt
  - Le Kremlin-Bicêtre
  - Lille
  - Montpellier
  - Nice
  - Paris
  - Rennes
  - Suresnes
- Germany (12):
  - Aachen
  - Bochum
  - Bonn
  - Frankfurt am Main
  - Halle
  - Hamburg
  - Jena
  - Kiel
  - Kÿln
  - Mainz
  - Marburg
  - Ulm
- Cork, Ireland
- Madrid, Spain
- Sweden (5):
  - Gothenburg
  - Huddinge
  - Linköpng N/A
  - Örebro
  - Stockholm
- Switzerland (4):
  - Geneva
  - Lucerne
  - Sankt Gallen
  - Zurich
- United Kingdom (4):
  - Edinburgh
  - London
  - N/a N/a
  - Salford

REFERENCES:
- [Result] Grond S, Hall J, Spacek A, Hoppenbrouwers M, Richarz U, Bonnet F. Iontophoretic transdermal system using fentanyl compared with patient-controlled intravenous analgesia using morphine for postoperative pain management. Br J Anaesth. 2007 Jun;98(6):806-15. doi: 10.1093/bja/aem102. PMID 17519263